CLINICAL TRIAL: NCT01015989
Title: Computerized Counseling to Promote Positive Prevention and HIV Health in Kenya
Acronym: CARE+ Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Indiana University (Other); Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH085577 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2018-09

CONDITIONS: HIV Infections
Keywords: HIV treatment; ART adherence; Using new technology to improve adherence; CARE+; HIV-1 viral loads
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Masking Description: The CARE Kenya counseling tool software randomizes the participant automatically to the control or intervention arms when the user first logs into the program, using a quasi-random number algorithm.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CARE+ Kenya brief computer risk assessment session (control) (Active Comparator)
  Interventions: Other: CARE+ Kenya brief computer risk assessment session
- Full CARE+ Spanish computer-counseling group (Active Comparator)
  Interventions: Other: CARE+ Kenya computer counseling session

INTERVENTIONS:
Other: CARE+ Kenya brief computer risk assessment session — The computer will ask patients questions about taking HIV medicine. The computer will also ask patients questions about sexual and substance use activities. We will repeat the session every 3 months up to 9 months total.
  Arms: CARE+ Kenya brief computer risk assessment session (control)
Other: CARE+ Kenya computer counseling session — The computer will ask patients questions about taking HIV medicine. The computer will also ask patients questions about sexual and substance use activities. The computer will let patients look at short videos on various HIV medicine and HIV risk reduction topics and will then help patients create a health plan. Patients will get an anonymous print out at the end of the session and can choose to share with health care provider. There are questions about depression, suicide, or domestic violence. If a patient's answers indicate that they may be depressed, suicidal, or currently in an abusive relationship, we will refer them to a health worker at the clinic. We will repeat the session every 3 months up to 9 months total.
  Arms: Full CARE+ Spanish computer-counseling group

SUMMARY:
The purpose of this study is to see if a computerized counseling tool helps patients reduce their sexual transmission risk and improve their antiretroviral adherence.

DETAILED DESCRIPTION:
Helping people living with HIV to remain healthy and reduce transmission to sexual partners ('positive prevention') can be accomplished by behavioral counseling and supporting adherence to infectivity-reducing antiretroviral therapy (ART). Positive prevention and ART adherence approaches that are not staff-dependent are urgently needed in Africa, the region hardest hit by HIV and decimated health workforce. Interactive health communication tools offer one approach. We will adapt a computerized counseling intervention found to be efficacious in reducing HIV-1 viral load and risk behaviors in the US ('CARE+') with the largest HIV provider in Kenya, the Academic Model for the Prevention and Treatment of HIV/AIDS (AMPATH). Aim 1: Adapt a theoretically driven computerized counseling intervention for use in Kenya ('CARE+_Kenya'). Conduct in-depth interviews with n≤ 50 urban and rural AMPATH patients to understand HIV support needs, and two staff focus groups to assess counseling practices and beliefs about computer use. Modify intervention content; translate and record audio into local Kiswahili. Adapt skill-building videos (e.g., on secondary prevention, HIV disclosure, ART adherence, reproductive health). Conduct software usability testing with n=20 patients and n=8 staff. Perform 3-day test-retest reliability assessment to establish psychometric performance of measures.

Aim 2: Establish biological and behavioral efficacy of CARE+_Kenya. Longitudinal randomized controlled trial (RCT) in one urban and one rural AMAPATH clinic. Randomly assign HIV-positive adults with any missed ART or unprotected sex in last 6 months, >1 sex partner in last year, or sexually transmitted infection (STI)diagnosis in last 3 years, to intervention (n=125) or risk-assessment control (n=125) for baseline, 3, 6, and 9 month sessions. HIV transmission risk will be measured by self-reported unprotected sex with HIV negative/unknown partner, and trends in Chlamydia trachomatis, Neisseria gonorrhoeae, and T. vaginalis. ART adherence will be measured by HIV-1 viral load, electronic monitoring, pharmacy refill, self-report, and clinic attendance. Aim 3: Establish cost-effectiveness of CARE+_Kenya. At baseline, follow 100 patients at each of the two clinics to evaluate standard of care counseling, and collect time-spent and facility data to determine costs and unmet counseling need. Conduct economic evaluation to compare CARE+_Kenya vs. standard of care. If the RCT shows that the intervention reduces viral load and transmission risk behaviors, we will use a Bernoulli transmission dynamics model to estimate number of secondary HIV infections prevented; then create a cost-effectiveness model to calculate 2 incremental cost-effectiveness ratios: 1) cost per HIV infection averted, and 2) cost per daily adjusted life year saved. If CARE+_Kenya is efficacious and efficient, we will develop a proposal for a cluster-randomized trial to assess translational effectiveness of CARE+_Kenya throughout the AMPATH system. This is directly responsive to PA-08-107's call for innovative, integrated interventions that leverage ART roll-out infrastructure in international settings to benefit people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Seen for care including ART at the clinics
* Able to understand spoken Kiswahili or English
* Reported less than "perfect" ART adherence/any missed dose or pill counts that indicate non-adherence with medication or delay in pharmacy refill; unprotected sex in the last 6 months, or >1 sex partner in last year, or any STI diagnosis in last 3 years
* Able to give consent (i.e., no evidence of inebriation or psychosis)

Exclusion Criteria:

* Not fluent in Kiswahili or English
* Has a thought disorder that precludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
ART adherence will be measured by HIV-1 viral load, electronic monitoring, pharmacy refill, self-report, and clinic attendance | Every 3 months up to 9 months
HIV transmission risk will be measured by self-reported unprotected sex with HIV negative/unknown partner, and trends in Chlamydia trachomatis, Neisseria gonorrhoeae, and T. vaginalis. | Every 3 months up to 9 months
We will conduct economic evaluation to compare CARE+ Kenya vs. standard of care. | 9 months

SECONDARY OUTCOMES:
Qualitative exit interviews with patients | At end of study
Two focus groups with providers | At end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kurth, PhD, Principal Investigator — NYU
Locations (2):
- Kenya (2):
  - AMPATH at Burnt Forest Health Centre, Burnt Forest, Rift Valley
  - AMPATH Module 1, Eldoret